CLINICAL TRIAL: NCT01124227
Title: Symptomatic Improvement by Peritoneal Dialysis in Patients With End Stage Congestive Heart Failure
Brief Title: Peritoneal Dialysis in Congestive Heart Failure
Acronym: PDinCHF
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to very specific inclusion criteria the anticipated number of patients was not reached. Inclusion stopped at N=26, allowing for analyzing primary outcomes.
Sponsor: Martini Hospital Groningen (Other)
Collaborators: Baxter Healthcare Corporation (Industry); Roche BV Netherlands (Unknown)
Responsible Party: Principal Investigator, Wilbert Martien Theodoor Janssen, MD PhD, Martini Hospital Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PDinCHF; 2009-017711-15 (EudraCT Number)
Record Dates: First submitted 2010-05-12; First posted 2010-05-17 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Congestive Heart Failure
Keywords: Congestive Heart Failure; Peritoneal Dialysis; Symptomatic improvement; Renal function
MeSH Terms: conditions — Heart Failure | interventions — Icodextrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard Care (Sham Comparator)
  Interventions: Drug: icodextrin
- 2 Icodextrin PD changes / day (Active Comparator)
  Interventions: Drug: icodextrin
- 1 Icodextrin PD change/day (Active Comparator)
  Interventions: Drug: icodextrin

INTERVENTIONS:
Drug: icodextrin — 2000 ml icodextrin intraperitoneally one or two times a day. Dose will be adapted clinically as in standard peritoneal dialysis.
  Other Names: Extraneal; RVG 21300

SUMMARY:
Rationale: End-stage congestive heart failure is a serious invalidating condition with a poor prognosis and increasing incidence. Non-randomized observations showed peritoneal dialysis (PD) in these patients to improve clinically from NYHA stadium III-IV to as low as NYHA stadium I-II. A randomized trial is needed to test whether PD improves symptoms in this condition and to find an optimal scheme.

Objective: To improve symptomatology in severe chronic failure patients. Study design: Open, parallel intervention trial comparing 2 schemes of peritoneal dialysis with icodextrin (Extraneal®) with standard medical therapy..

Study population: Patients with chronic refractory left ventricular congestive heart failure (LVEF < 30%, older than 18 years).

Intervention: Peritoneal dialysis with one (night) or two (night and day) dwells with icodextrin (Extraneal®).

Main study parameters/endpoints: Reduction in NYHA classification of symptomatic Congestive Heart Failure at 8 months after start of PD therapy. Burden of congestive heart failure: measured by reduction in unfavorable days (noted by patients in diaries and including days of hospitalization for CHF-deterioration and death).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Refractory Left Ventricular Congestive Heart Failure: LVEF < 30%
* Diminished renal function: eGFR < 60 ml/min
* Clinically volume overloaded (Dyspnoea (NYHA III-IV), edema, and/or ascites)
* Hospitalization for CHF during the last 6 months
* Patient is on optimal cardiologic medical therapy, which has been stable for more than 4 weeks
* Suitable for PD

Exclusion Criteria:

* Hypotension (SBP < 100 mmHg / MAP < 70) mmHg
* Instable AP or recent (< 6 months) myocardial infarction.
* Contraindications for PD (e.g. visual handicap, social)
* Liver failure
* COPD Gold class IV
* Malignancy with life expectancy < 2 years
* Non compliance
* No informed consent
* Poor mental health

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-04; Primary Completion 2016-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Number of patients in NYHA class I, II, III, or IV as measure of quality of life | 8 months

SECONDARY OUTCOMES:
Quality of life measures | 8 months
  Reduction in unfavorable days. Short-Form 36. Minnesota Living with Heart failure Questionnaire. 6 minute walk test. (re)hospitalization. Survival. Medication optimalisation. Cardial: LVH. Renal: GFR/ERPF/FF; KIM-1, NGAL, NAG. Volume status: ECV (radioactive and bio-impedance). Neurohumoral and inflammatory parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Wilbert M Janssen, MD, PhD, Principal Investigator — Martini Hospital
Locations (1):
- Martini Hospital, Groningen, Netherlands